CLINICAL TRIAL: NCT03777475
Title: the Effect of Different Oxaliplatin Dose in Transarterial Infusion (TAI) in Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong-ping Guo, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017-005-01
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose (Experimental): low oxaliplatin (85mg/m2)
  Interventions: Procedure: transarterial infusion
- high dose (Active Comparator): high oxaliplatin (135mg/m2)
  Interventions: Procedure: transarterial infusion

INTERVENTIONS:
Procedure: transarterial infusion — transarterial infusion

SUMMARY:
evaluate the effect of different oxaliplatin dose in TAI in treating unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old and younger than 75 years;
* ECOG PS≤1;
* proven hepatocellular carcinoma according patological examination or EASL/AASLD diagnostic criteria;
* not previous treated for tumor;
* unresectable;
* the lab test could meet: neutrophil count≥2.0×109/L; hemoglobin≥100g/L; platelet count≥75×109/L; serum albumin≥35g/L; total bilirubin<2-times upper limit of normal; ALT<3-times upper limit of normal; AST<3-times upper limit of normal; serum creatine<1.5-times upper limit of normal; PT≤upper limit of normal plus 4 seconds; INR≤2.2;
* sign up consent

Exclusion Criteria:

* cannot tolerate TAI or surgery;
* known history of other malignancy;
* be allergic to related drugs;
* underwent organ transplantation before;
* be treated before (interferon included);
* known history of HIV infection;
* known history of drug or alcohol abuse;
* have GI hemorrhage or cardiac/brain vascular events within 30 days;
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, assessed up to 60 months
  overall survival

SECONDARY OUTCOMES:
ORR | From date of randomization until the date of death from any cause, assessed up to 60 months
  object response rate
PFS | From date of randomization until the date of progress from any cause, assessed up to 60 months
  progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- SUN YAT-SEN University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided